CLINICAL TRIAL: NCT03358225
Title: A Muti-Center Study Comparing 3 Procedures for Bi-level Cervical Spondylosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Liu Haiying, department of spinal surgery, Peking University People's Hospital
Other Study IDs: Hybrid007
Record Dates: First submitted 2017-11-26; First posted 2017-11-30 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Cervical Spondylosis
Keywords: Hybrid surgery,ACDF,C-ADR,bi-level cervical spondylosis
MeSH Terms: conditions — Spondylosis | interventions — Gene Fusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Anterior Cervical Discectomy and Fusion: The patients undergoing anterior cervical discectomy and fusion surgery
  Interventions: Procedure: anterior cervical discectomy and fusion
- Cervical Artificial Disc Replacement: The patients undergoing cervical artificial disc replacement surgery
  Interventions: Procedure: cervical artificial disc replacement
- Hybrid surgery: The patients undergoing hybrid surgery(1-level ADR plus 1-level ACDF) surgery
  Interventions: Procedure: hybrid surgery

INTERVENTIONS:
Procedure: anterior cervical discectomy and fusion — The patients undergoing anterior cervical discectomy and fusion sugery
  Groups: Anterior Cervical Discectomy and Fusion
Procedure: cervical artificial disc replacement — The patients undergoing cervical artificial disc replacement surgery
  Groups: Cervical Artificial Disc Replacement
Procedure: hybrid surgery — The patients undergoing 1-level C-ADR plus 1-level ACDF surgery
  Groups: Hybrid surgery

SUMMARY:
A muti-center study to compare the safety and efficacy of anterior cervical discectomy and fusion, cervical artificial disc replacement and hybrid surgery for bi-level cervical spondylosis.

DETAILED DESCRIPTION:
Patients with bi-level cervical spondylosis undergoing anterior cervical discectomy and fusion, cervical artificial disc replacement and hybrid surgery in the muti-center hospital were retrospectively reviewed.The safety and efficacy were evaluated based on scores of the Neck Disability Index (NDI), visual analog scale (VAS), and Japanese Orthopedic Association (JOA) and the range of motion of both operative segments and adjacent segments,not only in the preoperative,but also in the 5 days,6 months,12 months and the 5 years after surgery.

ELIGIBILITY:
Inclusion Criteria:

* (1) Cervical degenerative pathology with symptomatic radiculopathy or myelopathy at two consecutive segments from C3 to C7 which not responding to conservative treatment for 6 weeks. (2) Preoperative magnetic resonance imaging (MRI), complete cervical spine radiography and computed tomography (CT) showed anterior compressive pathology. (3) None or slight osteophyte at the posterior edge of vertebrae. (4) None significant spinal stenosis or posterior compression.

Exclusion Criteria:

* ossification of the posterior longitudinal ligament (OPLL), tumor, fracture, infection, history of cervical spine surgery, narrowing of the spinal canal, and any serious general illness. Cases with one or more than two segments requiring treatment were also excluded.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with bi-level cervical spondylosis
Sampling Method: Non-Probability Sample
Enrollment: 198 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2018-12-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
range of the motion of operative segments and adjacent segments | preoperatively, within 5 days after surgery, and at 6, and 12 months postoperatively
  Standard dynamic flexion and extension lateral cervical radiographs were obtained to evaluate range of motion of C2-C7 and operative segments and superior and inferior adjacent segments, cervical lordosis, and radiographic changes in adjacent segments.

SECONDARY OUTCOMES:
scores of the Japanese Orthopedic Association | preoperatively, within 5 days after surgery, and at 6, and 12 months postoperatively
  Clinical effects were evaluated based on scores of the Japanese Orthopedic Association (JOA)
scores of the Neck Disability Index | preoperatively, within 5 days after surgery, and at 6, and 12 months postoperatively
  Clinical effects were evaluated based on scores of the Neck Disability Index(NDI)
scores of the visual analog scale | preoperatively, within 5 days after surgery, and at 6, and 12 months postoperatively
  Clinical effects were evaluated based on scores of the visual analog scale(VAS)

CONTACTS AND LOCATIONS:
Overall Officials: LIU Haiying, Principal Investigator — department of spinal surgery,PekingUPH

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Toledano M, Bartleson JD. Cervical spondylotic myelopathy. Neurol Clin. 2013 Feb;31(1):287-305. doi: 10.1016/j.ncl.2012.09.003. PMID 23186905
- [Background] Lebl DR, Hughes A, Cammisa FP Jr, O'Leary PF. Cervical spondylotic myelopathy: pathophysiology, clinical presentation, and treatment. HSS J. 2011 Jul;7(2):170-8. doi: 10.1007/s11420-011-9208-1. Epub 2011 Jun 22. PMID 22754419
- [Background] Veeravagu A, Cole T, Jiang B, Ratliff JK. Revision rates and complication incidence in single- and multilevel anterior cervical discectomy and fusion procedures: an administrative database study. Spine J. 2014 Jul 1;14(7):1125-31. doi: 10.1016/j.spinee.2013.07.474. Epub 2013 Oct 11. PMID 24126076
- [Background] Jia Z, Mo Z, Ding F, He Q, Fan Y, Ruan D. Hybrid surgery for multilevel cervical degenerative disc diseases: a systematic review of biomechanical and clinical evidence. Eur Spine J. 2014 Aug;23(8):1619-32. doi: 10.1007/s00586-014-3389-5. Epub 2014 Jun 8. PMID 24908252
- [Background] Lee MJ, Dumonski M, Phillips FM, Voronov LI, Renner SM, Carandang G, Havey RM, Patwardhan AG. Disc replacement adjacent to cervical fusion: a biomechanical comparison of hybrid construct versus two-level fusion. Spine (Phila Pa 1976). 2011 Nov 1;36(23):1932-9. doi: 10.1097/BRS.0b013e3181fc1aff. PMID 21289581